CLINICAL TRIAL: NCT00435344
Title: Provider and Peer Delivered Youth Smoking Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01CA080254-01A1 (NIH)
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2007-02-14 (Estimated); Status verified 2007-02

CONDITIONS: Tobacco Dependence
Keywords: Pediatric practice; Smoking cessation; Smoking prevention; Adolescents
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

INTERVENTIONS:
Behavioral: Pediatric Practice-Based Smoking Intervention

SUMMARY:
The purpose of this study was to determine whether a pediatric practice-based smoking prevention and cessation intervention increases abstinence rates among adolescents.

DETAILED DESCRIPTION:
The majority of adolescent smokers are interested in quitting and have attempted to stop with limited success. A recent review of cessation trials for adolescents has concluded that there are no proven programs to help teens stop smoking, but suggested interventions based on cognitive behavioral therapy and sensitive to stages of change appear promising. The American Academy of Pediatrics suggests that pediatricians are well-positioned to intervene with adolescent smokers, as well as with nonsmokers to prevent initiation. A comprehensive, practice-based smoking prevention and cessation intervention for adolescents delivered by pediatric providers and peer counselors in the context of routine care has the potential for assisting nonsmoking adolescents in remaining smoke-free and smoking adolescents to quit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 to 17, regardless of smoking status
* Scheduled for routine or acute care office visit
* Parental consent and youth assent

Exclusion Criteria:

* Unable to complete study requirements

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2711
Dates: Start 1999-02; Study Completion 2004-01

PRIMARY OUTCOMES:
Abstinence from smoking in the past 30 days at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, Ph.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Pbert L, Flint AJ, Fletcher KE, Young MH, Druker S, DiFranza JR. Effect of a pediatric practice-based smoking prevention and cessation intervention for adolescents: a randomized, controlled trial. Pediatrics. 2008 Apr;121(4):e738-47. doi: 10.1542/peds.2007-1029. PMID 18381502